CLINICAL TRIAL: NCT07307313
Title: Effectiveness of Motivational Interviewing Versus Traditional Patient Education in Promoting Oral Health Among Children
Brief Title: Effectiveness of Motivational Interviewing in Promoting Oral Health Among Children
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lamis D. Rajab (Other)
Responsible Party: Sponsor-Investigator, Lamis D. Rajab, professor, University of Jordan
Organization: University of Jordan (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UJordanLamis3
Record Dates: First submitted 2025-12-14; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Pediatric Dentistry; Motivational Interview, OHI; Motivational Intervention; Oral Hygiene Education Methods; Oral Hygiene, Oral Health
Keywords: Oral health; Oral hygiene; Clinical trial; video; Oral hygiene instructions; OHI; Oral hygiene education; Motivational interviewing; Traditional methods; Written instructions; Verbal instructions; Plaque score; Bleeding score
MeSH Terms: interventions — Videotape Recording

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Motivational interviewing (Experimental)
  Interventions: Behavioral: Motivational interviewing oral hygiene instructions
- Video (Experimental)
  Interventions: Other: Video for oral hygiene instructions
- Written and verbal instructions (Experimental)
  Interventions: Other: Written and verbal oral hygiene instructions

INTERVENTIONS:
Behavioral: Motivational interviewing oral hygiene instructions — Brief motivational interviewing session for each patient for around 20-30 minutes
  Arms: Motivational interviewing
Other: Video for oral hygiene instructions — A video about oral hygiene instructions uploaded from NHS and translated for the mother tongue language of the participants
  Arms: Video
Other: Written and verbal oral hygiene instructions — Basic oral hygiene instruction will be given verbally and then supported by written instructions.
  Arms: Written and verbal instructions

SUMMARY:
The goal of this clinical study is to compare the effect of motivational interviewing (MI) and traditional patient education methods in improving oral hygiene (plaque score and bleeding score) among young children 8-10. It will also assess the demographic (age and sex) and socioeconomic indicators' effect on oral hygiene (plaque score and bleeding score) after intervention.

The main questions this study aims to answer are:

* Is MI significantly more effective in improving oral health (plaque score, bleeding score) among children when compared to traditional patient education methods?
* Are there specific demographic or contextual factors (e.g., age, socioeconomic status, baseline oral health status) that influence the effectiveness of MI in promoting oral health among children when compared to traditional patient education methods?

Participants will be randomly assigned to three groups to receive oral hygiene instructions: verbal and written, video, and motivational interviewing.

Have their oral hygiene assessed using the plaque index and bleeding index before the intervention and after a follow-up period of 1 month.

DETAILED DESCRIPTION:
This clinical study aims to compare the effect of motivational interviewing (MI) and traditional patient education methods in improving oral hygiene (plaque score and bleeding score) among young children aged 8-10. The study is a randomized clinical trial that will be conducted among healthy pediatric patients attending the pediatric dentistry clinics at the University of Jordan Hospital.

Patients who meet the inclusion criteria and give consent will be randomly assigned to three groups:

1. Verbal and written instructions group: Basic oral hygiene instruction will be given to this group on a model of the mouth and then supported by written instructions.
2. Video monitored (VIDEO) group: Uploaded from the National Health Service (NHS) website and translated to the patient's mother tongue (Arabic).
3. Motivational interviewing (MI) group: The participants will join the motivation sessions one-to-one, face-to-face, with the primary researcher, who will be trained and calibrated to provide MI and take sessions with qualified psychologists.

Oral hygiene will be assessed using two parameters:

Plaque index scoring: 0/1 Bleeding on probing score: 0/1 Each patient will be examined twice: the first time is before the intervention, and the second is after a follow-up period of 1 month.

The study will also investigate the influence of age, sex, and socioeconomic status on oral hygiene improvement.

The findings of this research aim to contribute to the growing body of literature on MI and inform public health strategies aimed at reducing the global burden of childhood dental diseases.

ELIGIBILITY:
Inclusion Criteria:

* Children who are medically healthy
* Children with normal manual dexterity
* Children whose parents/guardians provide informed consent
* Children not currently receiving orthodontic therapy
* Children who do not require periodontal specialty care
* Children with normal occlusion or mild, non-treatment-requiring malocclusion

Exclusion Criteria:

* Children with systematic, or syndromic disease
* Children with special health care needs
* Children with poor manual dexterity
* Children with negative consents.
* Children with current orthodontic therapy
* Children with chronic diseases.
* Children on medications that may cause drug-induced gingivitis.
* Children who attend periodontal clinics.
* Children with malocclusion

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Plaque index | From enrollment to the 4-week follow-up appointment
  The primary researcher will document the plaque index for each patient prior to the intervention and after the follow-up appointment after 1 month using Plaque Control Index scoring
Bleeding index | From enrollment to the 4-week follow-up appointment
  The primary researcher will document the bleeding index for each patient prior to the intervention and during every follow-up appointment using Gingival Bleeding Index (GBI)

IPD SHARING:
Plan to Share IPD: Yes